CLINICAL TRIAL: NCT02780791
Title: Transplantation of Ovarian Tissue Into the Pelvic Wall and the Ovary After Cryopreservation of Ovarian Tissue Before Cytotoxic Therapies - Where do More Follicles Grow?
Brief Title: Maturation of Follicles After Transplantation of Ovarian Tissue Into the Pelvic Wall and the Ovary
Acronym: Ovartrans
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruited participants due to a lack of collaborating study centers
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-OVARTRANS
Record Dates: First submitted 2016-04-29; First posted 2016-05-23 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Infertility; Ovarian Failure, Premature
Keywords: Infertility; Ovarian Failure, Premature; Ovarian Follicle; Ovary; Tissue Transplantation; Cryopreservation; Pelvis; Chemotherapy; Pregnancy Rate; Folliculogenesis; Endometrium; Estrogens; Progestins; Follicle Stimulating Hormone; Estradiol; Progesterone; Hormones; Maturation of Follicles; Pregnant Women; Premature Menopause; Ovarian Insufficiency; Ovarian Insufficiency, Premature; Cytotoxic therapy; Fertility Protection; Reproductive Medicine; Reproductive Techniques; Reproductive Technology; Cryotherapy; Pregnancy
MeSH Terms: conditions — Infertility; Primary Ovarian Insufficiency; Menopause, Premature; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transplantation into pelvic wall (Active Comparator): Ovarian transplantation into the pelvic wall after cryopreservation of ovarian tissue before cytotoxic therapies
  Interventions: Other: Transplantation into pelvic wall
- Transplantation into the ovary (Active Comparator): Ovarian transplantation into ovary after cryopreservation of ovarian tissue before cytotoxic therapies
  Interventions: Other: Transplantation into the ovary

INTERVENTIONS:
Other: Transplantation into pelvic wall — Ovarian tissue will be transplanted subperitoneal into the loge of the adnexa of Uterus.
  Arms: Transplantation into pelvic wall
Other: Transplantation into the ovary — Ovarian tissue will be transplanted contralateral into the ovary.
  Arms: Transplantation into the ovary

SUMMARY:
The purpose of this study is to determine whether the pelvic wall or the ovary represents a better location for the maturation of follicles in the context of ovarian transplantation after cryopreservation of ovarian tissue before cytotoxic therapies.

DETAILED DESCRIPTION:
The development of modern medicine made it more likely for oncological patients to survive. Also, there are a lot of young female patients with a persistent wish for kids. After an aggressive chemotherapy, premature ovarian failure (POF) is a possible consequence of the therapy. Therefore, efficient fertility protective interventions are requested. The transplantation of ovarian tissue after cryopreservation is a valuable method, which could remain fertility after POF induced by cytotoxic therapies. Especially for girls suffering from cancer, who didn't reach puberty yet, cryopreservation of ovarian tissue is the only opportunity to preserve a chance of restoring fertility after POF.

There are two locations, which could be used for the retransplantation of the cryopreserved tissue: the remaining ovary and the pelvic wall. Both, the ovary and the subperitoneal pocket in the pelvic wall present a location, where the maturation of follicles is possible. The remaining question is: where do more follicles grow? To answer this question, a study will be necessary. The purpose of this study is to determine whether the pelvic wall or the ovary represents a better location for the maturation of follicles in the context of ovarian transplantation after cryopreservation of ovarian tissue before cytotoxic therapies.

Interventions:

Ovarian tissue will be transplanted into two different locations; subperitoneal into the loge of the adnexa of uterus and contralateral into the ovary. The assignment of the two parts of ovarian tissue to the place of transplantation (pelvic wall vs. ovary) will be randomised. The study-specific interventions include:

* Transplantation of the same amount of ovarian tissue into both locations
* Monthly sonographic controls and determination of estradiol, LH, FSH and progesterone from the 3rd on to the 12th month after the transplantation. Therefore, blood samples will be made.
* Monthly documentation of the duration of the cycle from the 3rd on to the 12th month after transplantation

One year after the transplantation, the investigators will be able to determine which location is more likely to grow follicles. With the gained knowledge, standardized recommendations could be formulated which help to improve the whole process of medical care of female oncologist patients.

ELIGIBILITY:
Inclusion Criteria:

* Age at cryopreservation ot tissue max. 38 years
* Age at transplantation 18-49 years
* At least one maintained ovary
* Premature ovarian failure
* Indication for an autologous transplantation of ovarian tissue
* Permitted pregnancy from the part of the oncologists
* Written informed consent

Exclusion Criteria:

* Age at transplantation <18 and >49 years
* Cryopreservation in the context of a leucaemia, neuroblastoma, Burkitt-lymphoma

Important: Inclusion is only done by one of the recruiting centers. Study participation will only be given on invitation. Please contact Principal Investigator!

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2017-09-10 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Comparison of follicle maturation in transplanted tissue between pelvic wall and ovary | Beginning 3 months after the transplantation until 12 months after the transplantation
  The participants will get an assessment of the follicle maturation on both sides (pelvic wall and ovary) each month beginning 3 months after the transplantation until 12 months after the transplantation. Overall, 10 assessments will take place. The maturation of follicles will be detected with sonography and measured in mm.
  Along with the sonography, blood samples will be taken and examined for their amount of estradiol, FSH and progesterone. A follicle ≥15mm with a concentration of estradiol >500 pmol/L (>136pg/ml) is considered a mature follicle.
  The primary outcome contains the quantitative comparison of mature follicles grown on both sides.

SECONDARY OUTCOMES:
Duration of cycle, measured in weeks | Beginning 3 months after the transplantation until 12 months after the transplantation
  The participants will be asked for the duration of their last cycle (2, 3, 4, 5, 6, 7, 8 weeks or no cycle). The assessments will take place monthly, beginning 3 months after the transplantation until 12 months after the transplantation.
Number of study participants with pregnancy | 12 months after transplantation and 24 months after transplantation
  Documentation of pregnancy ratio after transplantation of autologous ovarian tissue
Number of study participants with life-birth after pregnancy | 12 months after transplantation and 24 months after transplantation
  Documentation of life-birth ratio after pregnancy in context after transplantation of autologous ovarian tissue
Determination of hormone levels after transplantation, concerning the concentration of estradiol, progesterone, LH, FSH | Beginning 3 months after the transplantation until 12 months after the transplantation
  Blood samples will be examined for their amount of estradiol, progesterone, FSH and LH in order to check the vitality and the functionality of the transplanted tissue.
Sonographic measurement of the endometrium wall, measured in mm | Beginning 3 months after the transplantation until 12 months after the transplantation
  Monthly sonographic measurement of the endometrium wall will be performed. Along with the determination of hormone levels after the transplantation, these measurements hold a more detailed evaluation of the activity of the transplanted tissue and his effect on a functional organ (e.g. endometrium).

CONTACTS AND LOCATIONS:
Overall Officials: Michael von Wolff, Prof.Dr.med., Principal Investigator — Universitätsfrauenklinik, Abteilung für Gynäkologische Endokrinologie und Reproduktionsmedizin, Effingerstrasse 102, 3010 Bern
Locations (1):
- Universitätsfrauenklinik, Abteilung für Gynäkologische Endokrinologie und Reproduktionsmedizin, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The Source data will include:
  * All documents required in the Trial master file
  * Visit dates and participation in the study along with consent forms
  * Completed CRFs and patient medical charts
  * All documentation related to SAEs and AEs
  * All documentation related to concomitant medication and results of study relevant examinations
  Direct access to source documents will be permitted for purposes of monitoring, audits and inspections. Access to protocol, dataset, statistical code during and after the study will be given to the PI, the other defined investigators, the persons who perform the monitoring and the statistician.
  The key to decode the health related data will be stored at the Universitätsfrauenklinik, Abteilung Gynäkologische Endokrinologie und Reproduktionsmedizin, Effingerstrasse 102, 3010 Bern. The access to the key will only be given to persons, who need it to fulfill their tasks in the sense of the study.